CLINICAL TRIAL: NCT03639740
Title: TReat-to-tArget (T2T) With seCukinumab in Axial Spondyloarthritis. IdEntification of MRI and Biochemical Biomarkers for Disease Activity, Treatment Response and Structural Damage Progression (the TRACE Study)
Brief Title: Treat-to-target With Secukinumab in Axial Spondyloarthritis
Acronym: TRACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Professor Mikkel Østergaard (Other)
Collaborators: Novartis Healthcare A/S (Industry)
Responsible Party: Sponsor-Investigator, Professor Mikkel Østergaard, Professor, DMSc, PhD, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TRACE; 2017-004037-93 (EudraCT Number)
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Axial Spondyloarthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Dose will be increased or maintained after predetermined intervals depending on remission
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Secukinumab 150 mg 300 mg or tumor necrosis factor inhibitor (Other): Secukinumab 150 mg sc. injection once a week for four weeks (induction phase) and thereafter once a month. If patients do not achieve ASDAS remission they get increased dosage of Secukinumab 300 mg sc. injection once a month. If still no ASDAS remission patients change to a TNF-inhibitor
  Interventions: Drug: Secukinumab 150 milligram [Cosentyx]

INTERVENTIONS:
Drug: Secukinumab 150 milligram [Cosentyx] — For intervention description: see arm/group description
  Other Names: Secukinumab 300 milligram [Cosentyx]

SUMMARY:
A study of axSpA and AS receiving Secukinumab in a treat-to-target strategy.

DETAILED DESCRIPTION:
Comparison of reductions in MRI inflammation in the sacroiliac joints and spine from week 16 to 24 in patients who at week 16 are in ASDAS remission (i.e. continue sc. secukinumab 150 mg monthly) vs. not in ASDAS remission (i.e. increase sc. secukinumab 300 mg monthly). ASDAS remission is defined as ASDAS inactive disease i.e. ASDAS<1.3.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of axial spondyloarthritis (axSpA) according to the ASAS (Assessment of Spondyloarthritis International Society) criteria and/or ankylosing spondylitis (AS) according to the modified New York criteria as judged by a spondyloarthritis (SpA) rheumatologist (regarding imaging in the criteria, see below).
2. Active inflammation on MRI of the SIJs and/or spine as evaluated by a central SpA imaging expert and/or radiographic modified New York criteria fulfilled as judged by a central SpA imaging expert.
3. Active disease defined as ASDAS ≥ 2.1 (ASDAS high disease activity).
4. Total back pain as measured on a visual analogue scale (VAS) scale ≥ 4 0 mm (0-100 mm) at baseline.
5. Clinical indication for a biologic drug as assessed by the treating physician.
6. Patients should have received at least 2 different NSAIDs at the highest recommended dose for at least 2 weeks each with an inadequate response or failure to respond, or less if therapy had to be reduced due to intolerance, toxicity or contraindications.
7. Patients on NSAIDs at inclusion should stay on a stable dose from at least 2 weeks before the baseline MRI scans are performed and to the week 24 visit.
8. Patients on synthetic disease-modifying anti-rheumatic drugs (sDMARDs) at inclusion should stay on a stable dose from at least 4 weeks before initiation of secukinumab to the week 24 visit.
9. Patient must be able to understand and communicate with the investigator and comply with the requirements of the study and must provide written, signed and dated informed consent before any study assessment is performed.
10. Male or female patients at least 18 years and less than 70 years of age.
11. Sufficient contraception for women.
12. Age ≥18 to <70 years.
13. Capable of giving informed consent.
14. Capable of complying with the examination programme of the protocol.

Exclusion Criteria:

1. Contraindications for secukinumab (described in protocol).
2. Contraindication for TNF inhibitor (described in protocol).
3. Contraindication for MRI (described in protocol).
4. Previous exposure to secukinumab or other biologic drug directly targeting interleukin-17 or interleukin-17 receptor.
5. Previous exposure to TNF inhibitor or drug targeting TNF.
6. Previous exposure to other types of biological disease-modifying anti-rheumatic drugs (bDMARDs) than TNF inhibitor.
7. Patients taking high-potency opioid analgesics (e.g. methadone, hydromorphone, morphine)
8. Any change in the dose of oral corticosteroids in the last 8 weeks prior to the baseline visit or use of i.v. intramuscular or intra-articular corticosteroid during the last 8 weeks prior to the enrollment visit.
9. Use of any investigational drug and/or devices within 4 weeks before randomization or a period of 5 half-lives of the investigational drug, whichever is longer.
10. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
11. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during the entire study or longer if required by locally approved prescribing information (e.g. 20 weeks in EU).
12. Known recent drug or alcohol abuse.
13. Incapable of complying with the examination programme for physical or mental reasons.
14. Failure to provide written consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a positive change in MRI-inflammation | Comparison of week 16 and 24
  Assessed with the sum of SPARCC MRI SIJ and spine inflammation indices

SECONDARY OUTCOMES:
Proportion of patients in remission vs patients not in ASDAS (Ankylosing Spondylitis Disease Activity Score) remission. | Comparison of week 16 and 24
  as measured by remission (<1.3) / not in ASDAS remission (>1.3)
Changes in ASDAS score (i.e. Ankylosing Spondylitis Disease Activity Score (ASDAS 0.6-7.0)) | Evaluated from week 0 to 16 and from week 16 to 24
  as measured by changes in ASDAS.
Changes in MRI inflammation scores from week 0 to 16 and week 16 to 24, respectively. | Week 0 to 16 and week 16 to 24
  as measured by the SPARCC MRI SIJ and Spine Inflammation indices and the Canada-Denmark MRI system for a positive change in MRI inflammation in the spine as assessed with the Canada-Denmark MRI system for assessment of inflammation.
Changes in scores/anatomical location of MRI lesions in the spine | week 16
  as measured by the Canada-Denmark MRI system for assessment of inflammation, fat metaplasia, erosion, and new bone formation.
Changes in scores/anatomical location of MRI lesions in the SIJs | week 16
  as measured by the SPARCC MRI SIJ Inflammation Index and SPARCC SIJ Structural Score (SSS)
MRI inflammation | week 16
  as measured by the SPARCC (Spondyloarthritis Research Consortium of Canada) MRI sacroiliac joint and Spine Inflammation indices and the Canada-Denmark MRI system for assessment of inflammation assessed on cMRI (conventional MRI) i.e. on STIR (short tau inversion recovery) sequences on conventional and novel scan planes and on DWI (Diffusion-weighted imaging) sequences evaluated visually and based on regions of interest (ROIs).

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Østergaard, DMSc PhD MD, Principal Investigator — Rigshospitalet, Denmark; Susanne J Pedersen, MD PhD, Study Chair — Rigshospitalet, Denmark
Locations (10):
- Denmark (10):
  - Reumatologisk Afdeling, Aarhus Universitetshospital, Aarhus
  - Videncenter for Reumatologi og Rygsygdomme, Rigshospitalet - Frederiksberg, Frederiksberg
  - Videncenter for Reumatologi og Rygsygdomme, Rigshospitalet Glostrup, Glostrup Municipality
  - Kong Christian X´s Gigthospital, Gråsten
  - Videncenter for Reumatologi og Rygsygdomme, Rigshospitalet - Gentofte, Hellerup
  - Videncenter for Reumatologi og Rygsygdomme, Rigshospitalet - Nordsjællands Hospital Hillerød, Hillerød
  - Reumatologisk Afdeling, Regionshospitalet Nordjylland, Hjørring, Hjørring
  - Reumatologisk afdeling, Sjællands Universitetshospital, Køge, Køge
  - Reumatologisk Afdeling, Odense Universitetshospital, Odense
  - Reumatologisk Afdeling, Regionshospitalet Silkeborg, Silkeborg